CLINICAL TRIAL: NCT05324228
Title: Determination of Reference Values for Sublingual Microcirculation in Healthy Volunteers in the Pediatric Population Using the Sidestream Dark-Field Imaging Method
Brief Title: Sublingual Microcirculation in Healthy Children Using the SDF Imaging Method
Status: Completed | Type: Observational
Sponsor: Vlasta Krausová (Other)
Responsible Party: Sponsor-Investigator, Vlasta Krausová, Principal Investigator, Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s.
Organization: Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s. (Other)
Other Study IDs: 300/7
Record Dates: First submitted 2022-03-27; First posted 2022-04-12 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Healthy
Keywords: Microcirculation; Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Preschool children: 10 preschool healthy children aged 3-5,9 years.
- Children of younger school age: 10 children of younger school age aged 6-10,9 years.
- Children in puberty: 10 children in puberty aged 11-14,9 years
- Postpubertal adolescents: 10 postpubertal adolescents aged 15-18,9 years.

SUMMARY:
The main goal of the study is to determine the physiological parameters of sublingual microcirculation in children in different age categories using Sidestream Dark-Field Imaging Method. No significant differences are expected to be found between measurements in healthy volunteers in different age categories.

DETAILED DESCRIPTION:
After recording the basic anthropometric parameters, pressure, pulse and O2 saturation, each volunteer who meets the inclusion criteria will have their microcirculation measured using a Sidestream Dark-Field (SDF) probe placed sublingually by one examiner using the SDF method. The measurement will be performed in supine position in a disease-free period, with normal diets, at least 2 hours after the last meal in the afternoon, for girls outside the menses period. Premedication or analgesia will not be used. A total of 3 video clips will be recorded from different parts of the sublingual area with a minimum length of 20 seconds in a row, unless the child needs a short break between measurements. The recorded videos will then be processed offline by one evaluator who is trained and experienced in microcirculation evaluation, three best and most stable parts of each video clip will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* healthy child
* informed consent of parents

Exclusion Criteria:

* inability to cooperate
* acute illness
* chronic illness
* chronic medication
* substance abuse

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will include 40 healthy volunteers. Of these, 10 pre-school children (3-5.9 years), 10 younger school children (6-10.9 years), 10 children in puberty(11-14.9 years) and 10 post-puberty adolescents will be included (15-18.9 years).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Determination of Total Vascular Density of sublingual microcirculation of children | baseline
  Total length of vessels divided by total surface of area
Determination of Microvascular Flow Index (MFI) of sublingual microcirculation of children | baseline
  The image is divided into four quadrants and the predominant type of flow (absent = 0, intermittent = 1, sluggish = 2, normal = 3, and hyperdynamic = 4) is assessed in each quadrant. The MFI score represents the averaged values of the four. A 20 μm cut-off is used to separate small vessels (mostly capillaries) from large vessels (mostly venules).
Determination of Small Vessel Density of sublingual microcirculation of children | baseline
  Total length of small vessels divided by total surface of area. A 20 μm cut-off is used to separate small vessels (mostly capillaries) from large vessels (mostly venules).
Determination of Proportion of Perfused Vessels (all) of sublingual microcirculation of children | baseline
  The proportion of perfused vessels (PPV [%]) can be calculated as follows: 100 × (total number of vessels - [no flow + intermittent flow])/total number of vessels.
Determination of Proportion of Perfused Small Vessels (PPV) of sublingual microcirculation of children | baseline
  The proportion of perfused small vessels (PPV [%]) can be calculated as follows: 100 × (total number of small vessels - [no flow + intermittent flow])/total number of small vessels.
  A 20 μm cut-off is used to separate small vessels (mostly capillaries) from large vessels (mostly venules).
Determination of Perfused Vessel Density (all) of sublingual microcirculation of children | baseline
  Total length of vessels - (no flow + intermittent flow) divided by total surface of area
Determination of Perfused Small Vessel Density (PVD) of sublingual microcirculation of children | baseline
  Total length of small vessels - (small vessels with no flow + intermittent flow) divided by total surface of area. A 20 μm cut-off is used to separate small vessels (mostly capillaries) from large vessels (mostly venules).
Determination of DeBacker Score of sublingual microcirculation of children | baseline
  In this score, three equidistant horizontal and three equidistant vertical lines are drawn on the screen. Vessel density can be calculated as the number of vessels crossing the lines divided by the total length of the lines.

SECONDARY OUTCOMES:
Differences in Total Vascular Density in children of different age categories | baseline
  Total length of vessels divided by total surface of area. Comparison in children aged 3-5,9; 6-10,9; 11-14,9; and 15-18,9 years.
Differences in Microvascular Flow Index (MFI) in children of different age categories | baseline
  The image is divided into four quadrants and the predominant type of flow (absent = 0, intermittent = 1, sluggish = 2, normal = 3, and hyperdynamic = 4) is assessed in each quadrant. The MFI score represents the averaged values of the four. A 20 μm cut-off is used to separate small vessels (mostly capillaries) from large vessels (mostly venules). Comparison in children aged 3-5,9; 6-10,9; 11-14,9; and 15-18,9 years.
Differences in Small Vessel Density in children of different age categories | baseline
  Total length of small vessels divided by total surface of area. A 20 μm cut-off is used to separate small vessels (mostly capillaries) from large vessels (mostly venules).Comparison in children aged 3-5,9; 6-10,9; 11-14,9; and 15-18,9 years.
Differences in Proportion of Perfused Vessels (all) in children of different age categories | baseline
  The proportion of perfused vessels (PPV [%]) can be calculated as follows: 100 × (total number of vessels - [no flow + intermittent flow])/total number of vessels. Comparison in children aged 3-5,9; 6-10,9; 11-14,9; and 15-18,9 years.
Differences in Perfused Vessel Density (all) in children of different age categories | baseline
  Total length of vessels - (no flow + intermittent flow) divided by total surface of area. Comparison in children aged 3-5,9; 6-10,9; 11-14,9; and 15-18,9 years.
Differences in Proportion of Perfused Small Vessels (PPV) in children of different age categories | baseline
  The proportion of perfused small vessels (PPV [%]) can be calculated as follows: 100 × (total number of small vessels - [no flow + intermittent flow])/total number of small vessels.
  A 20 μm cut-off is used to separate small vessels (mostly capillaries) from large vessels (mostly venules). Comparison in children aged 3-5,9; 6-10,9; 11-14,9; and 15-18,9 years.
Differences in Perfused Small Vessel Density (PVD) in children of different age categories | baseline
  Total length of small vessels - (small vessels with no flow + intermittent flow) divided by total surface of area. A 20 μm cut-off is used to separate small vessels (mostly capillaries) from large vessels (mostly venules).Comparison in children aged 3-5,9; 6-10,9; 11-14,9; and 15-18,9 years.
Differences in DeBacker Score in children of different age categories | baseline
  In this score, three equidistant horizontal and three equidistant vertical lines are drawn on the screen. Vessel density can be calculated as the number of vessels crossing the lines divided by the total length of the lines. Comparison in children aged 3-5,9; 6-10,9; 11-14,9; and 15-18,9 years.

CONTACTS AND LOCATIONS:
Overall Officials: David Neumann, MD, Ph.D, Study Chair — University Hospital in Hradec Kralove
Locations (1):
- Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s., Ústí nad Labem, Czechia

IPD SHARING:
Plan to Share IPD: No